CLINICAL TRIAL: NCT04309136
Title: The Efficacy and Safety of Anlotinib in Neoadjuvant Treatment in Locally Advanced Thyroid Cancer: a Single-arm Phase II Clinical Trial
Brief Title: Anlotinib Neoadjuvant Treatment in Locally Advanced Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHNATHY
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; locally advanced; neoadjuvant; Anlotinib
MeSH Terms: conditions — Thyroid Neoplasms | interventions — anlotinib; Surgical Procedures, Operative; Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Anlotinib (Experimental)
  Interventions: Drug: Anlotinib; Procedure: surgery; Procedure: core needle biopsy

INTERVENTIONS:
Drug: Anlotinib — All patients will receive Anlotinib for at least two cycles of neoadjuvant treatment
Procedure: surgery — Perform surgery if operable after neoadjuvant therapy
Procedure: core needle biopsy — Perform core needle biopsy if inoperable after neoadjuvant therapy

SUMMARY:
To determine the efficacy and safety of Anlotinib in patients of locally advanced thyroid cancer in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteered to participate in the study and signed an informed consent form;
* Pathologically diagnosed locally advanced thyroid cancer, including papillary thyroid cancer, medullary cancer, follicular cancer, poorly differentiated cancer, etc., require surgical resection with or without distant metastasis;
* Preoperative assessment of invasion or adhesion of at least one of the following structures / organs, including: trachea, esophagus, common carotid artery, larynx, anterior vertebral fascia, brachial plexus, intended for surgical treatment;
* Have at least one measurable lesion (RECIST 1.1);
* Age 14-80 years, Eastern Cooperative Oncology Group (ECOG) score 0-1;
* The main organ functions meet the following criteria within 7 days before treatment:

  1. Standard blood test (without blood transfusion within 14 days):Hemoglobin (HB) ≥90g / L;Absolute neutrophil value (ANC) ≥ 1.5 × 109 / L;Platelet (PLT) ≥80 × 109 / L
  2. Biochemical inspection must meet the following standards:Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN, if with liver metastases, ALT and AST ≤ 5 ULN; Serum creatinine (Cr) ≤ 1.5 ULN or creatinine clearance (CCr) ≥ 60ml / min;
  3. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).
* Women of childbearing age should agree to use contraceptives during the study and within 6 months after the study; negative serum or urine pregnancy tests within 7 days before study enrollment; men should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Previously used anlotinib or similar VEGFR-TKI small molecule drugs, such as vandetanib, cabozantinib, lenvatinib, sunitinib, sorafenib and etc.
* Received external radiation therapy or iodine-131 therapy within the past 3 months; or planned systemic anti-tumor therapy during this study;
* Pathologically confirmed non-thyroid epithelial cell-derived malignant tumors (including lymphoma, metastatic cancer, sarcoma, etc.);
* With other uncontrolled / under treatment malignancies;
* Those who have multiple factors (such as inability to swallow) that affect oral medication;
* With pleural effusion or ascites, causing respiratory syndrome (≥CTC AE level 2 dyspnea [level 2 dyspnea refers to shortness of breath when a small amount of activity; affecting instrumental daily activities]);
* Patients with any severe and / or uncontrolled illness, including:

  1. Patients whose blood pressure is still unsatisfactory with a blood pressure medication (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg);
  2. Patients with myocardial ischemia or myocardial infarction of grade I or higher and congestive heart failure of grade 2 or higher (New York Heart Association (NYHA) classification);
  3. Sinus bradycardia; or atrioventricular block of more than two degrees, or sinus arrest (except for pacemakers); arrhythmia (including QTC ≥480ms); need to be used together to extend QTc interval drugs, including those for antiarrhythmic treatment;
  4. Active or uncontrolled severe infection (≥CTC AE level 2 infection);
  5. Patients with cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis;
  6. Renal failure requires hemodialysis or peritoneal dialysis;
  7. Have a history of immunodeficiency, including those who are HIV positive or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
  8. Poor blood glucose control in diabetic patients (fasting blood glucose (FBG)> 10mmol / L);
  9. Urine routine indicates urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g.
* received major surgical treatment, incisional biopsy or obvious traumatic injury within 28 days before enrollment;
* Patients whose imaging showed that the tumor had invaded the important blood vessels or the researchers judged that the tumor was likely to invade important blood vessels during the subsequent study period and caused fatal bleeding;
* Patients with any signs or history of bleeding regardless of severity; patients with any bleeding or bleeding event ≥ CTCAE level 3 within 4 weeks prior to grouping with unhealed wounds, ulcers or fractures
* Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism within 6 months;
* History of aneurysm;
* Those with a history of epilepsy or neurological disorders with ataxia in need of treatment;
* People with a history of psychotropic substance abuse who are unable to quit or have mental disorders;
* Those with a history of peripheral nervous system disease and muscle strength below 3;
* Those who have participated in other clinical trials of anti-tumor drugs within four weeks or are conducting other clinical trials;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of patients or affect patients to complete the research.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at the time point of 18 weeks
  ORR

SECONDARY OUTCOMES:
R0/1 resection rate | at the time of surgery
  R0/1 resection rate if operable
Disease control rate | at the time point of 18 weeks
  DCR
Overall survival | up to 3 years
  OS
Adverse Events | from the first drug administration to within 90 days after surgery
  AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang NS, Wei WJ, Xiang J, Chen JY, Guan Q, Lu ZW, Ma B, Sun GH, Wang YL, Ji QH, Wang Y. The Efficacy and Safety of Anlotinib in Neoadjuvant Treatment of Locally Advanced Thyroid Cancer: A Single-Arm Phase II Clinical Trial. Thyroid. 2021 Dec;31(12):1808-1813. doi: 10.1089/thy.2021.0307. Epub 2021 Nov 29. PMID 34610756